CLINICAL TRIAL: NCT03659448
Title: Multicenter, Open-label, Randomized, Controlled, Parallel Arms Clinical Study on Performance of SGM-101, a Fluorochrome-labeled Anti-CEA Monoclonal Antibody, for Delineation of Primary/Recurrent Tumor and Metastases in Patients Undergoing Surgery for Colorectal Cancer
Brief Title: Performance of SGM-101 for the Delineation of Primary and Recurrent Tumor and Metastases in Patients Undergoing Surgery for Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Surgimab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SGM-CLIN03
Record Dates: First submitted 2018-05-04; First posted 2018-09-06 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Neoplasms
Keywords: Fluorescence; Cancer; SGM-101; Surgery; Colorectal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Two parallel arms consisting of a treatment arm of patients who will receive the study drug and subsequently undergo surgical resections under both "standard "white light" conditions and then NIR, and a no treatment arm to whom the study drug will not be administered and who will undergo surgical resections under standard "white light" conditions only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Patients will receive a single dose of the study drug, SGM-101, and subsequently undergo surgical resections under both "standard "white light" conditions and then NIR.
  Interventions: Drug: SGM-101
- No Treatment (No Intervention): Patients will not be administered the study drug, SGM-101, and will undergo surgical resections under standard :white light" conditions only.

INTERVENTIONS:
Drug: SGM-101 — A fluorochrome-labeled anti-carcinoembryonic antigen (CEA) monoclonal antibody intraoperative imaging agent.
  Arms: Treatment

SUMMARY:
The performance of SGM-101, an intraoperative imaging agent, will be compared to that of standard "white light" visualization during surgical resections of colorectal cancer.

DETAILED DESCRIPTION:
The performance of SGM-101, a fluorochrome-labeled anti-carcinoembryonic antigen (CEA) monoclonal antibody intraoperative imaging agent for the delineation of primary and recurrent tumor and metastases in patients undergoing curative surgery for colorectal cancer will be compared to that of standard "white light" visualization in a multicenter, open-label, randomized, controlled, parallel arms clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be scheduled for curative colorectal cancer surgery of primary cT4 colon cancer or primary cT3/4 rectal cancer, recurrent colorectal cancer or peritoneal metastasized colorectal cancer.
* Female patients must be of non-child-bearing potential (i.e., women with functioning ovaries who have a documented tubal ligation or hysterectomy, ovariectomy or women who are post-menopausal). Women of child-bearing potential will be included provided that they have a negative urine pregnancy test at the day of the injection and agree to practice adequate contraception for 30 days prior to administration of investigational product, and 30 days after completion of injection.

Exclusion Criteria:

1. Other malignancies, either currently active or diagnosed in the last 5 years, except for adequately treated in situ carcinoma of the cervix and basal or squamous cell skin carcinoma;
2. Primary appendiceal cancer;
3. Laboratory abnormalities defined as:

   * Aspartate AminoTransferase, Alanine AminoTransferase, Gamma Glutamyl Transferase) or Alkaline Phosphatase levels above 5 times the ULN or;
   * Total bilirubin above 2 times the ULN or;
   * Serum creatinine above 1.5 times the ULN or;
   * Absolute neutrophils counts below 1.5 x 109/L or;
   * Platelet count below 100 x 109/L or;
   * Hemoglobin below 4 mmol/L (females) or below 5 mmol/l (males);
4. Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody or patients with untreated serious infections;
5. Any condition that the investigator considers to be potentially jeopardizing the patient's well-being or the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Surgical resection histopathology. | Through completion of surgery, up to 9 weeks.
  Comparison of surgical resections using histopathology as standard of truth..

CONTACTS AND LOCATIONS:
Overall Officials: Alex L. Vahrmeijer,, MD, PhD, Principal Investigator — Leiden University Medical Center, Leiden, The Netherlands
Locations (11):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Moores Cancer Center - UCSD Health, La Jolla, California
  - Cleveland Clinic Florida, Weston, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
- Universitätsmedizin Göttingen, Klinik für Allgemein- Viszeral- und Kinderchirurgie, Göttingen, Germany
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy
- Netherlands (3):
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Leiden University Medical Center, Leiden
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No